CLINICAL TRIAL: NCT00652431
Title: SCH 465981: Assessment of Bi-Directional Interaction Between Components of Vytorin® (Ezetimibe and Simvastatin) and Niaspan® (Niacin Extended-Release Tablets) in Healthy Subjects
Brief Title: Assessment of Interaction Between Vytorin and Niaspan in Healthy Subjects (P04955AM2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P04955; Doc ID: 3498819
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Hyperlipidemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — Ezetimibe, Simvastatin Drug Combination; Niacin; Ezetimibe; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vytorin + Niaspan (Experimental): NIASPAN 1000 mg (1 x 1000 mg tablet) once-daily in the morning on Days 1 to 2, followed by NIASPAN 2000 mg (2 x 1000 mg tablets) once-daily in the morning on Days 3 to 7 + VYTORIN 10/20 mg (1 x 10/20 mg tablet containing ezetimibe 10 mg and simvastatin 20 mg) once-daily in the morning for 7 days
  Interventions: Drug: Vytorin + Niaspan
- Vytorin (Active Comparator): VYTORIN 10/20 mg (1 x 10/20 mg tablet containing ezetimibe 10 mg and simvastatin 20 mg) once-daily in the morning for 7 days
  Interventions: Drug: Vytorin
- Niaspan (Active Comparator): NIASPAN 1000 mg (1 x 1000 mg tablet) once-daily in the morning on Days 1 to 2, followed by NIASPAN 2000 mg (2 x 1000 mg tablets) once-daily in the morning on Days 3 to 7 for a total of 7 days of treatment
  Interventions: Drug: Niaspan

INTERVENTIONS:
Drug: Vytorin + Niaspan — Vytorin (1 tablet containing ezetimibe 10 mg and simvastatin 20 mg) once daily in the morning for 7 days + Niaspan 1000 mg (1 x 1000-mg tablet) once daily in the morning on Days 1 and 2, followed by Niaspan 2000 mg (2 x 1000-mg tablets) once daily in the morning on Days 3 to 7
  Other Names: SCH 465981; ezetimibe; simvastatin; niacin; nicotinic acid
  Arms: Vytorin + Niaspan
Drug: Vytorin — Vytorin (1 tablet containing ezetimibe 10 mg and simvastatin 20 mg) once daily in the morning for 7 days
  Other Names: SCH 465981; ezetimibe; simvastatin
  Arms: Vytorin
Drug: Niaspan — Niaspan 1000 mg (1 x 1000-mg tablet) once daily in the morning on Days 1 and 2, followed by Niaspan 2000 mg (2 x 1000-mg tablets) once daily in the morning on Days 3 to 7
  Other Names: niacin; nicotinic acid
  Arms: Niaspan

SUMMARY:
This is a single-center, randomized, open-label, 3-period, 3-treatment multiple-dose crossover study designed to assess the interaction between VYTORIN® (Ezetimibe and Simvastatin) and NIASPAN® (Niacin Extended-Release Tablets) in healthy subjects. Treatment spans 7 days

ELIGIBILITY:
Inclusion Criteria:

The subject must meet ALL the criteria listed below for entry:

* Subjects must be willing to give written informed consent and able to adhere to dose and visit schedules.
* Subjects of either sex and of any race between the ages of 18 and 55 years, inclusive, having a Body Mass Index (BMI) between 19 to 32, inclusive. BMI = weight (kg)/height (m^2).
* Subjects' clinical laboratory tests (CBC, blood chemistry, and urinalysis) must be within normal limits or clinically acceptable to the investigator/sponsor. Subject's liver function test results (AST, ALT, and GGT) must not be elevated above normal limits at Screening and on Day-1. Subjects' CPK test results must not be elevated more than 1.25 times the upper limit of normal, at Screening and on Day -1.
* Subjects must be free of any clinically significant disease that would interfere with the study evaluations.
* Screening ECG conduction intervals must be within gender specific normal range (QTc males <=430 msec and females <=450 msec).
* Vital sign measurements (taken after ~3 minutes in a seated position) must be within the following ranges:

  * oral body temperature between 35.0°C to 37.5°C
  * systolic blood pressure, 90 to 140 mm Hg
  * diastolic blood pressure, 45 to 90 mm Hg
  * pulse rate, 40 to 100 bpm
* Female subjects of childbearing potential must have a negative serum pregnancy test (beta-hCG) at Screening and have a negative urine pregnancy test upon each admission to the study center.
* Women of child-bearing potential must agree to use medically accepted methods of contraception prior to screening, while receiving protocol-specified medication, and for 30 days after stopping the medication. Acceptable methods of contraception include:

  * Condoms (male or female) with spermicide,
  * Diaphragm or cervical cap with spermicide
  * Medically prescribed IUD with spermicide, and
  * Surgical sterilization (eg. hysterectomy or tubal ligation). Vasectomy of the partner should be considered a single barrier and one additional contraceptive methods listed above must be used. Females who are not currently sexually active must agree and consent to use one of the above-mentioned methods should they become sexually active while participating in the study.
* Female subjects must be surgically sterilized (eg, documented hysterectomy or tubal ligation) or be postmenopausal. (Defined as 12 months with no menses and with an estradiol level of <30 pg/mL.)
* Men must agree to use a medically accepted method of contraception prior to Screening, while receiving protocol-specified medication, and for 30 days after stopping the medication.

Exclusion Criteria:

The subject will be excluded from entry if ANY of the criteria listed below are met:

* Female subjects who are pregnant, intend to become pregnant (within 3 months of ending the study), or are breastfeeding.
* Subjects who, in the opinion of the investigator, will not be able to participate optimally in the study.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug. The investigator should be guided by evidence of any of the following and be discussed with the sponsor prior to enrollment into the trial:

  * history or presence of inflammatory bowel disease, ulcers, gastrointestinal or rectal bleeding;
  * history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
  * history of pancreatic injury or pancreatitis;
  * history or presence of liver disease or liver injury;
  * history or presence of impaired renal function as indicated by abnormal creatinine, urinary albumin, BUN/urea or clinical significant urinary cellular constituents (eg, cast); or
  * history of urinary obstruction or difficulty in voiding.
* Subject who has a history of any infectious disease within 4 weeks prior to drug administration.
* Subjects who are positive for hepatitis B surface antigen, hepatitis C antibodies or HIV.
* Subjects who have a positive screen for drugs with a high potential for abuse.
* Subjects with a history of mental instability or who have been treated for mood disorders.
* Subjects with a history of alcohol or drug abuse in the past 2 years.
* Subjects who have donated blood in the past 60 days.
* Subjects who have previously received and demonstrated intolerance to NIASPAN® (niacin extended-release tablets), VYTORIN® (ezetimibe/simvastatin), ZETIA® (ezetimibe), ZOCOR® (simvastatin) or products containing niacin/nicotinic acid.
* Subjects who are currently participating in another clinical study or have participated in a clinical study within 30 days.
* Subjects who are part of the study staff personnel or family members of the study staff personnel.
* Subjects who have demonstrated allergic reactions (eg, food, drug, atopic reactions or asthmatic episodes).
* Subjects who smoke more than 10 cigarettes or equivalent tobacco use per day.
* Subjects who have received any treatment listed in Table 2 of protocol P04955 (Doc ID: 3498819) more recently than the indicated washout period prior to Baseline in each period.
* Subjects who received vaccination(s) within 30 days prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the potential for a PK interaction between NIASPAN and components of VYTORIN, using Tmax, Cmax, and AUC. | Day 7

SECONDARY OUTCOMES:
Evaluate safety and tolerability: laboratory test results, ECGs, adverse events, vital signs. | throughout study

REFERENCES:
- [Result] Kosoglou T, Zhu Y, Statkevich P, Triantafyllou I, Taggart W, Xuan F, Kim KT, Cutler DL. Assessment of potential pharmacokinetic interactions of ezetimibe/simvastatin and extended-release niacin tablets in healthy subjects. Eur J Clin Pharmacol. 2011 May;67(5):483-92. doi: 10.1007/s00228-010-0955-6. Epub 2010 Dec 1. PMID 21120461